CLINICAL TRIAL: NCT06979388
Title: A Phase I, Randomised, Single-dose, Open-label, 3-period, 3-treatment, 3-way Crossover Study to Assess the Effect of Food on Balcinrenone/Dapagliflozin Pharmacokinetics in Fed and Fasted State and Pharmacokinetics of Balcinrenone When Dosed With a P-gp Inhibitor in Healthy Participants.
Brief Title: A Study to Investigate the Effect of Food on Balcinrenone/Dapagliflozin Pharmacokinetics in Fed and Fasted State and Pharmacokinetics of Balcinrenone When Dosed With a P-gp Inhibitor in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6402C00009; 1011789 (Other: IRAS)
Record Dates: First submitted 2025-05-05; First posted 2025-05-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Food effect; Mineralocorticoid receptor modulator; P-glycoprotein inhibitor; Fed and fasted state; Standardised high-fat and high-calorie meal
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency; Fasting | interventions — dapagliflozin; Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment ABC (Experimental): Participants will receive Treatment A (reference, fasted), balcinrenone/dapagliflozin capsule on Day 1 and then followed by a washout period of 72 hours. On Day 4, participants will receive Treatment B (fed), balcinrenone/dapagliflozin capsule dosed together with food, followed by a washout period of 72 hours. On Day 7, participants will receive Treatment C (quinidine, fasted), balcinrenone/dapagliflozin capsule dosed together with a P-gp inhibitor tablets (2 doses of quinidine separated by 4 hours, 1 hour prior and 3 hours post balcinrenone/dapagliflozin administration, respectively).
  Interventions: Drug: balcinrenone/ dapagliflozin; Drug: quinidine
- Treatment ACB (Experimental): The participants will receive Treatment A (reference, fasted), balcinrenone/dapagliflozin capsule on Day 1 and then followed by washout period of 72 hours. On Day 4, participants will receive Treatment C (quinidine, fasted), balcinrenone/dapagliflozin capsule dosed together with a P-gp inhibitor tablets (2 doses of quinidine separated by 4 hours, 1 hour prior and 3 hours post balcinrenone/dapagliflozin administration, respectively), followed by a washout period of 72 hours. On Day 7, participants will receive Treatment B (fed), balcinrenone/dapagliflozin capsule dosed together with food.
  Interventions: Drug: balcinrenone/ dapagliflozin; Drug: quinidine
- Treatment BCA (Experimental): The participants will receive Treatment B (fed), balcinrenone/dapagliflozin capsule dosed together with food on Day 1 and then followed by washout period of 72 hours. On Day 4, participants will receive Treatment C (quinidine, fasted), balcinrenone/dapagliflozin capsule dosed together with a P-gp inhibitor tablets (2 doses of quinidine separated by 4 hours, 1 hour prior and 3 hours post balcinrenone/dapagliflozin administration, respectively), followed by a washout period of 72 hours. On Day 7, participants will receive Treatment A (reference, fasted), balcinrenone/dapagliflozin capsule.
  Interventions: Drug: balcinrenone/ dapagliflozin; Drug: quinidine
- Treatment BAC (Experimental): The participants will receive Treatment B (fed), balcinrenone/dapagliflozin capsule dosed together with food on Day 1 and then followed by washout period of 72 hours. On Day 4, participants will receive Treatment A (reference, fasted), balcinrenone/dapagliflozin capsule and then followed by washout period of 72 hours. On Day 7 participants will receive Treatment C (quinidine, fasted), balcinrenone/dapagliflozin capsule dosed together with a P-gp inhibitor tablets (2 doses of quinidine separated by 4 hours, 1 hour prior and 3 hours post balcinrenone/dapagliflozin administration, respectively).
  Interventions: Drug: balcinrenone/ dapagliflozin; Drug: quinidine
- Treatment CAB (Experimental): The participants will receive Treatment C (quinidine, fasted), balcinrenone/dapagliflozin capsule dosed together with a P-gp inhibitor tablets (2 doses of quinidine separated by 4 hours, 1 hour prior and 3 hours post balcinrenone/dapagliflozin administration, respectively), followed by a washout period of 72 hours. On Day 4, participants will receive Treatment A (reference, fasted), balcinrenone/dapagliflozin capsule and then followed by washout period of 72 hours. On Day 7, participants will receive Treatment B (fed), balcinrenone/dapagliflozin capsule dosed together with food.
  Interventions: Drug: balcinrenone/ dapagliflozin; Drug: quinidine
- Treatment CBA (Experimental): The participants will receive Treatment C (quinidine, fasted), balcinrenone/dapagliflozin capsule dosed together with a P-gp inhibitor tablets (2 doses of quinidine separated by 4 hours, 1 hour prior and 3 hours post balcinrenone/dapagliflozin administration, respectively), followed by a washout period of 72 hours. On Day 4, participants will receive Treatment B (fed), balcinrenone/dapagliflozin capsule dosed together with food, followed by a washout period of 72 hours. On Day 7, participants will receive Treatment A (reference, fasted), balcinrenone/dapagliflozin capsule.
  Interventions: Drug: balcinrenone/ dapagliflozin; Drug: quinidine

INTERVENTIONS:
Drug: balcinrenone/ dapagliflozin — Participants will be receiving balcinrenone/ dapagliflozine in fasted or fed condition.
Drug: quinidine — Participants will be receiving quinidine orally in fasted condition.

SUMMARY:
The main purpose of this study is to assess the effect of food on balcinrenone/ dapagliflozin pharmacokinetics in fed and fasted state and pharmacokinetics of balcinrenone when dosed with a P-gp inhibitor in healthy participants.

DETAILED DESCRIPTION:
This study will be an open-label, randomised, 3-period, 3-treatment, single-dose, 3-way crossover study in healthy participants (males and females), performed at a single study site.

The study comprises of:

* Screening period of 4 weeks within the interval of Day -28 and Day -2.
* Three treatment periods during which participants will be residing at the Clinical Unit from the day before the first study intervention administration (Day -1). The participant will be discharged on Day 10.

  * Treatment A (reference, fasted), balcinrenone/dapagliflozin capsule dosed in the fasted state.
  * Treatment B (fed), balcinrenone/dapagliflozin capsule dosed together with food.
  * Treatment C (quinidine, fasted), balcinrenone/dapagliflozin capsule (dosed together with a P-gp inhibitor tablets (quinidine) in fasted state.

Participants will be randomised on Day 1 to one of the following 6 treatment sequences: ABC, ACB, BCA, BAC, CAB, or CBA. Each participant will receive all 3 treatments (A, B, and C) in the sequence participant was randomised to. Each treatment will be separated by a washout period of 72 hours; thus, each participant will receive study intervention on Day 1, Day 4, and Day 7.

• A final Follow-up Call within 5 - 7 days (Day 12-14) after the last study intervention administration.

ELIGIBILITY:
Main Inclusion Criteria:

* Have a Body Mass Index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* All females of childbearing potential must have a negative pregnancy test.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception.

Main Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/major surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any clinically important abnormalities in clinical chemistry, haematology, urinalysis or vital signs.
* Positive result for serum hepatitis B surface antigen, hepatitis C antibody, and HIV antibody
* History of long QT syndrome or history of additional risk factors for QT prolongation - for example a family history of long QT syndrome or the use of concomitant medications known to prolong the QT/QTc interval. Any clinically significant abnormalities on 12-lead ECG at the Screening Visit, as judged by the investigator, including but not limited to any significant arrythmia, conduction abnormalities, and/or prolonged QTcF > 450 ms.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months prior to Screening Visit.
* History of alcohol or drug abuse. Positive screen for drugs of abuse, alcohol or cotinine.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* History of hypersensitivity to drugs with a similar chemical structure or class to balcinrenone, dapagliflozin and quinidine. Any contraindications listed for dapagliflozin and quinidine.
* Use of drugs with enzyme inducing properties within 3 weeks prior to the first administration of study intervention.
* Use of any prescribed or nonprescribed medication, herbal remedies or intake of > 3 × daily recommended levels of vitamins and minerals during the 2 weeks prior to the first administration of study intervention
* Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve from time zero to infinity (AUCinf) | From Day 1 to Day 10
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | From Day 1 to Day 10
Maximum observed drug concentration (Cmax) | From Day 1 to Day 10
Terminal elimination half-life (t1/2λz) | From Day 1 to Day 10
Time to reach maximum observed concentration (tmax) | From Day 1 to Day 10
Apparent volume of distribution based on the terminal phase (Vz/F) | From Day 1 to Day 10
Apparent total body clearance (CL/F) | From Day 1 to Day 10
Renal Clearance (CLR) (balcinrenone only) | From Day 1 to Day 10
Drug concentration in plasma at 24 hours post-dose (C24) | From Day 1 to Day 10

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From Screening (Day -28 to Day -2) until Follow-up (Day 12 to Day 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/